CLINICAL TRIAL: NCT01621724
Title: WT1 TCR Gene Therapy for Leukaemia: A Phase I/II Safety and Toxicity Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Medica Ltd (Industry)
Collaborators: University College, London (Other); Cell Therapy Catapult (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-00272-CT2014001
Record Dates: First submitted 2012-03-22; First posted 2012-06-18 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukaemia; Chronic Myeloid Leukaemia
Keywords: Gene therapy; WT1 TCR; AML; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm cohort study (Experimental): WT1 TCR-transduced T cells
  Interventions: Genetic: WT1 TCR-transduced T cells

INTERVENTIONS:
Genetic: WT1 TCR-transduced T cells — Two patient cohorts:
  Cohort 1 (up to 6 patients) = ≤ 2 x 107/kg WT1 TCR-transduced T cells
  Cohort 2 (12 patients)= ≤ 108/kg WT1 TCR-transduced T cells

SUMMARY:
WT1 TCR gene therapy is a new treatment for acute myeloid leukaemia and chronic myeloid leukaemia.

Patient's white blood cells (T cells) are modified to specifically fight the leukaemia cells by transferring a gene into the T cells, which allows them to recognize fragments of a protein called WT1. This protein is present on the surface of leukaemia cells at very high levels. The gene transferred to the T cells enables them to make a new T cell receptor (TCR), which will allow them to attack leukaemia cells with high levels of WT1 on their surface.

Using this form of gene therapy the investigators can convert some of the patient's immune system's own T cells into T cells that the investigators hope will be much more effective at recognizing and killing leukaemia cells.

DETAILED DESCRIPTION:
This trial concerns a novel approach to generating leukaemia antigen-specific T cells for adoptive cellular therapy in HLA-A*0201 patients with acute myeloid leukaemia (AML) and chronic myeloid leukaemia (CML)

In this study, patient T cells will be gene-modified using a GMP grade retroviral vector containing the genes for a WT1-specific, HLA-A2-restricted T cell receptor. This ex vivo gene therapy will generate T cells expressing the WT1-specific TCR and thus able to recognise WT1-expressing target cells.

The autologous Cys1 WT1 TCR-transduced T cells will be re-infused back into adult leukaemia patients following lymphodepleting conditioning.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Life expectancy ≥ 16 weeks (4 months).
* World Health Organisation (WHO) performance status of 0-2
* HLA A*0201 positive
* Completed previous course of chemotherapy ≥ 4 weeks prior to commencing the initial phase of the trial (leucapheresis for collection of patient PBMC).
* Peripheral blood total lymphocyte count > 0.5x109/L.
* Informed consent in writing and ability to co-operate with treatment and follow up.
* Willing, able and available for collection of PBMC/ T cells by leucapheresis.
* Hepatitis B and C, HTLV-1, Syphilis, HIV negative.
* Free from serious concurrent illness.
* Female patients of child-bearing age must have a negative pregnancy test and agree to use reliable contraceptive methods for the duration of the therapy and for 6 months afterwards.
* Male patients must agree to use appropriate medically approved contraception during the trial and for six months afterwards.
* Haematological and Biochemical Indices:
* Haemoglobin (Hb) ≥ 7.0 g/dl; neutrophils ≥ 0.2 x 109/L; total lymphocytes > 0.5 x 109/L; platelets (Plts) ≥ 40 x 109/L
* serum bilirubin, Alanine amino-transferase (ALT) and/or aspartate amino transferase (AST) < 3 x upper normal limit
* calculated creatinine clearance ≥ 30 ml/min (uncorrected value) or isotope clearance measurement ≥ 30ml/min

Further disease specific inclusion criteria are detailed in Protocol

Exclusion Criteria:

* Age < 18 years or > 75 years.
* Patients should not receive concurrent systemic corticosteroids whilst on the study.
* Within three months of having received fludarabine (at time of leucapheresis).
* Major thoracic and/or abdominal surgery in the preceding three to four weeks from which the patient has not yet recovered.
* Patients who are high medical risks because of non-malignant systemic disease, as well as those with active uncontrolled infection.
* Patients with any other condition, which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Patients known to be serologically positive for Hepatitis B, C, HTLV-1 Syphilis or HIV.
* Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/ IV cardiac disease
* Positive pregnancy test or reluctance to use contraception.
* Pregnant and lactating women are excluded.
* History of Severe Allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Identify organ toxicities and other side effects | Up to 12 months per patient
Transduction efficiency and TCR expression on TCR-transduced cells | Up to 12 months per patient

SECONDARY OUTCOMES:
WT1-specific immune responses of TCR-transduced T cells | Up to 12 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Emma Morris, Dr, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University College London Hospitals NHS Trust, London